CLINICAL TRIAL: NCT06388291
Title: Double Blind Comparison of Optimised Deep Brain Stimulation for Severe Tourette Syndrome
Brief Title: Deep Brain Stimulation in Tourette Syndrome
Acronym: Op-TICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University College London Hospitals (Other); Northern Care Alliance NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); University of Bristol (Other); University of Dundee (Other); London School of Hygiene and Tropical Medicine (Other); King's College London (Other); University Hospital, Rouen (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CTU/2018/321
Record Dates: First submitted 2022-06-08; First posted 2024-04-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Tourette Syndrome; Deep Brain Stimulation
Keywords: Movement Disorders; Nervous System Diseases; Brain Diseases; Functional Disorder
MeSH Terms: conditions — Tourette Syndrome; Movement Disorders; Nervous System Diseases; Brain Diseases | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will have electrodes implanted in the globus pallidus interna and connected to a subcutaneous pulse generator.
  This will be followed by a 6 months open-phase period of stimulation for electrical parameter adjustment.
  Following these 6 months, participants will be randomised into two groups by the order of treatment condition (ON/OFF-stimulation vs OFF/ON-stimulation): for up to two weeks in each condition. Tic severity will be assessed and all participants will enter a 2-day interval, in the ON state, before switching to the other treatment condition for another two weeks.
  A mechanistic part of the study will look at possible explanations of differing responses in both the open and randomised phase. To identify the factors which predict the degree of response to DBS in TS the investigators will be looking at the role of: clinical factors: age, disease duration, tic severity at baseline, co-morbidity, Electrical parameters of stimulation, & Imaging.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ON/OFF-stimulation (Experimental): This group will have the stimulator switched on for two weeks followed by off for two weeks
  Interventions: Device: Deep Brain Stimulation
- OFF/ ON -stimulation (Experimental): This group will have the stimulator switched off for two weeks followed by on for two weeks
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — ON/OFF stimulation vs OFF/ON stimulation

SUMMARY:
Op-TICS is a clinical investigation of the use of Deep Brain Stimulation (DBS), with a CE marked implantable device, to reduce severe motor and vocal tics in patients who suffer from Tourette Syndrome (TS).

It is a randomised, double-blind, crossover clinical investigation for 20 patients. Op-TICS will be performed at the National Hospital for Neurology & Neurosurgery.

Following DBS surgery, participants will first enter an open adjustment phase, of 6 months, where the electrical stimulation settings of the device are optimised. Participants will then enter the double-blind phase that will include successively up to 2 weeks with stimulation on and up to 2 weeks with the stimulation off in a randomised order.

The primary outcome measure is the tic severity score measured by the Yale Global Tic Severity Scale -Total Tic Score after two weeks OFF-stimulation versus two weeks ON-stimulation in the double-blind randomised crossover phase

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a neuropsychiatric disorder with patients exhibiting multiple motor tics and at least one vocal tic. When these tics are distressing, medications or behavioural therapy can be used to control symptoms.

However, there are a small number of patients with very severe tics who are unresponsive to these conventional treatments and suffer a major negative impact on their quality of life. This limits their social interaction and access to most jobs. These patients are in urgent need of more effective treatments.

Deep brain stimulation (DBS) is a technique that involves the surgical implantation of two thin wires (electrodes) in the right and left globus pallidus, areas of the brain responsible for the control of body movement. The electrodes are connected to a stimulator placed on the chest under the skin that sends electrical signals to the brain. This type of surgery is routinely used for disorders such as Parkinson's disease and has also been used in a smaller number of TS patients.

DBS is an accepted treatment for conditions such as Parkinson's disease, dystonia and tremor. In experienced teams the risks associated with the surgery and the device are very low. A small number of patients with Tourette syndrome around the world have benefited from DBS; nevertheless, more evidence is needed before DBS can be made available as an NHS treatment for severely affected patients and NHS England has prioritised this research topic.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18 and over:

1. with chronic, severe, treatment refractory Tourette Syndrome, as defined by a Yale Global Tic Severity Scale score (YGTSS (global)) >50/100
2. with failure to respond to a minimum of two antipsychotic drugs prescribed separately at maximally tolerated doses for a minimum of 6 weeks OR, intolerance of these medications causing early cessation due to adverse events
3. who have provided agreement to participate and written informed consent

Exclusion Criteria:

1. Schizophrenia or other primary psychotic disorder (schizophrenia (ICD11 6A20); delusional disorders (ICD11 6A24); schizoaffective disorder (ICD11 6A21).
2. History of substance-induced psychotic disorder (ICD11 6C40.6 Alcohol-induced psychotic disorder; ICD11 6C43.6 Opioid-induced psychotic disorder; ICD11 6C41.6 Cannabis-induced psychotic disorder; ICD11 6C42.6 Synthetic cannabinoid-induced psychotic disorder; ICD11 6C44.6 Sedative, hypnotic or anxiolytic-induced psychotic disorder; ICD11 6C45.6 Cocaine-induced psychotic disorder; ICD11 6C46.6 Stimulant-induced psychotic disorder including amphetamines, methamphetamine or methcathinone; ICD11 6C47.6 Synthetic cathinone-induced psychotic disorder; 6C49.5 Hallucinogen-induced psychotic disorder; ICD11 6C4B.6 Volatile inhalant-induced psychotic disorder; ICD11 6C4C.6 MDMA or related drug-induced psychotic disorder, including MDA; ICD11 6C4D.5 Dissociative drug-induced psychotic disorder including Ketamine or PCP; ICD11 6C4E.6 Psychotic disorder induced by other specified psychoactive substance).
3. Recurrent depressive disorder with a history of attempted suicide (ICD11 6A71).
4. Bipolar disorder (ICD11 6A60).
5. Severe personality disorder judged to be contributing to impaired social function by the physician reviewing eligibility (ICD11 6D10.2).
6. Disorders of Intellectual Development (defined as moderate intellectual disabilities (ICD11 6A00.1); severe intellectual disabilities (ICD11 6A00.2); profound intellectual disabilities (ICD11 6A00.3)).
7. Autism Spectrum Disorders with exception of ICD11 6A02.0 Autism spectrum disorder without disorder of intellectual development and with mild or no impairment of functional language.
8. Significant cognitive impairment as judged at the discretion of the physician reviewing eligibility.
9. Pregnancy or absence of an acceptable method of contraception.
10. Contraindications to neurosurgery (such as brain abnormalities, haemostasis disorder or contraindication to MRI) or anaesthesia.
11. Severe intercurrent pathology and any other disease that could interfere with the protocol or compromise life expectancy, in the Investigator's judgement.
12. Continued participation in any other interventional clinical trials.
13. Any other implanted electronic devices such as implantable cardioverter defibrillators (ICD), permanent pacemakers (PPM) and drug pumps.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Tic severity score measured by the YGTSS-TTS (total tic) after two weeks OFF-stimulation versus two weeks ON-stimulation in the double-blind randomised crossover phase | 4 weeks
  To assess whether GPi DBS is effective in reducing severe motor or vocal tics, measured with the Yale Global Tic Severity Scale -Total Tic Severity (YGTSS- TTS) two weeks OFF stimulation vs two weeks ON Stimulation at the end of the double blind randomised crossover blinded phase, i.e., Effect 1 (Visit 5) vs Effect 2 (Visit 7)

SECONDARY OUTCOMES:
MRVRS at the end of the OFF-stimulation state versus the end of the ON-stimulation state in the blinded, randomised crossover phase. | 4 weeks
  TIC number and severity measured using the Modified Rush Video Rating Scale (MRVRS) at the end of the OFF-stimulation state (Visit 5) versus the end of the ON-stimulation state (Visit 7) in the blinded randomised phase
Change in the MRVRS between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  TIC number and severity measured using the MRVRS at Baseline 0 and Baseline 1
Change in the YGTSS (global) between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  TIC number, severity and complexity measured using the YGTSS at Baseline 0 and Baseline 1
Change in the GTS-QOL questionnaire measures at baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  Quality of life measured using the Gilles de la Tourette Syndrome - Quality Of Life (GTS-QoL) questionnaire at baseline 0 and baseline 1
Change in the YBOCS between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  Severity of obsessions and compulsions measured using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) at baseline 0 and baseline 1
Change in the BDI scale between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  Severity of depression measured using Beck Depression Index (BDI) at baseline 0 and baseline 1
Change in the BAI scale between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  Severity of anxiety measured using the Beck Anxiety Index (BAI) at baseline 0 and baseline 1
Change in the BAARS-IV between baseline 0 and the end of the open-phase (Baseline 1) | 24 weeks
  Severity of ADHD symptoms and domains of impairment measured using the Barkley Adult ADHD Rating Scale-IV (BAARS-IV) at baseline 0 and baseline 1
Safety of DBS as indicated by the number of participants with any adverse events and number with any serious adverse events | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of Neurology & Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No